CLINICAL TRIAL: NCT02995434
Title: Immersive Multimedia as an Adjunctive Measure for Pain Control in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other); Simon Fraser University (Other); Fraser Health (Other)
Responsible Party: Principal Investigator, Bernie Garrett, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H16-01510
Record Dates: First submitted 2016-10-12; First posted 2016-12-16 (Estimated); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain; Cancer
Keywords: Virtual Reality; Cancer Survivorship; Pain Management; Cancer Pain Management; Chronic Pain Management; Adjunctive Pain Management
MeSH Terms: conditions — Chronic Pain; Neoplasms; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will be randomly assigned to the intervention group (50 in total).The VR intervention will be identical for each participant and consist of a PC running the immersive virtual reality application with a Virtual Reality headset 110 degrees field of view head mounted display. The VR will be a set of commercial exploratory virtual environment games designed for the HTC Vive headset. The intervention will be used for one month to enable customization to the therapy and record data over a long enough period of time to account for individual short- term changes in pain experience. Participants will be asked to use the VR therapy every day with a time exposure of 30 minutes for four consecutive weeks. There will be one rest day a week (normally a Sunday) where no therapy is given.
  Interventions: Device: Virtual Reality Headset
- Control Group (Active Comparator): The control group will be exposed to 2D PC equivalent versions of the same multimedia experiences but on their PC screen (without the Virtual Reality headset use). These will be functionally similar to the VR experiences.
  Interventions: Other: 2D PC

INTERVENTIONS:
Device: Virtual Reality Headset — The following VR experiences will be used:
  Virtual Meditative Walk: http://painstudieslab.com/projects/virtual-meditative-walk/ Wildflowers: https://appadvice.com/app/wildflowers-mindfulness/988835763 Obduction: http://obduction.com/ Carpe Lucem: http://store.steampowered.com/app/433700/Carpe_Lucem__Seize_The_Light_VR/
  Other Names: HTC Vive
  Arms: Intervention Group
Other: 2D PC — The control group will be exposed to 2D equivalent versions of the same multimedia experiences but on their PC screen (without the VR headset use). These will be functionally similar to the VR experiences. These will include:
  Virtual Meditative Walk: http://painstudieslab.com/projects/virtual-meditative-walk/ Wildflowers: https://appadvice.com/app/wildflowers-mindfulness/988835763 Obduction: http://obduction.com/ The Witness: http://store.steampowered.com/app/210970/
  Arms: Control Group

SUMMARY:
This study seeks to explore the efficacy of immersive multimedia experiences as a practical adjunctive therapeutic intervention in the self-management of the chronic pain associated with cancer patients. A comparative controlled interventional trial and qualitative interpretative-descriptive exploration will be undertaken with 100 cancer patients who are experiencing chronic pain. Participants will be randomly assigned to either a virtual reality (VR) therapy group or a 2D computer based multimedia control group (50 subjects in each).

They will undertake either a series of VR interventions, or 2D computer based multimedia control sessions in their own homes over a period of a month. The intervention will be used daily for a month to enable customization to the therapy and record data over a long enough period of time to account for any individual short-term changes in pain.

The VR sessions will consist of using a VR head mounted display (HMD) and computer to explore interactive immersive environments. The control group will be exposed to similar 2D computer based multimedia experiences (without a VR headset) that on home computers. Pre, during, and post pain test scores and quality of sleep assessments will be recorded using standardized tools.

In addition to the primary study, a sub-study will be conducted where ten of the subjects who demonstrated the most improvement in their pain using the VR experience will be selected and invited to explore for any measurable changes in neurological activity using pre and post exposure electroencephalography (EEG).

DETAILED DESCRIPTION:
This study seeks to explore the efficacy of an immersive multimedia experience as a practical therapeutic intervention in the self-management of the chronic pain associated with cancer patients.

This work will inform further clinical studies and future research into the potential uses of immersive multimedia in the treatment of cancer associated pain. Furthermore, it will help identify optimal immersive multimedia environments for use in chronic pain applications, practical determinants for implementation of immersive multimedia for wider practice, and will provide a better theoretical understanding of the mechanisms whereby immersive multimedia works in chronic pain.

JUSTIFICATION

Cancer survivorship refers to individuals who have remained cancer free for a minimum of 5 years. Due to developments and greater outcomes associated with cancer therapy and management, the number of individuals who survive cancer has risen considerably over the past decade. Currently, 65% of adults and 80% of children can be expected to live at least 5 years post cancer diagnosis. However, for some, survivorship is associated with debilitating chronic pain which impacts negatively on quality of life. Reviews have suggested that up to 40% of individuals have survived cancer remain with cancer related chronic pain.

With rapidly emerging immersive multimedia technologies and clinical work in this field, it would appear that immersive multimedia may have significant potential for use as an adjunctive therapeutic measure for pain control. However, there has been little work done to establish the potential use of immersive multimedia in the management of chronic cancer pain to date, as most work on immersive multimedia for pain management has focused on acute pain via distraction. Several researchers have recommended the investigation of immersive multimedia for chronic, long term pain, and the research team completed a pilot study in 2015 to establish best methods and approaches for using immersive multimedia in chronic pain conditions.

OBJECTIVES

To determine if immersive multimedia therapy is effective as an adjunctive intervention in the management of chronic pain in cancer patients?

1. Can exposure to a immersive multimedia environment as an adjunctive pain-relieving measure provide a pain-reducing experience for for chronic cancer pain patients?
2. How long (if at all) do any therapeutic effects of immersive multimedia last after exposure in chronic cancer pain patients?
3. Are there any significant side effects of immersive multimedia exposure for chronic cancer pain patients?
4. Do any identifiable neurological changes occur on EEG pre and post immersive multimedia exposure?

RESEARCH METHODS

A longitudinal mixed-methods study to evaluate the impact of immersive multimedia for chronic pain in cancer patients is proposed which will consist of a comparative controlled interventional trial and qualitative interpretative-descriptive exploration.

1. Interventional Trial (Quantitative):

   Participants will be randomly assigned to either a VR therapy group or the control group (50 subjects in each). They will undertake either a series of immersive VR interventions, or control sessions (using 2D multimedia on personal computers) in their own homes over a period of a month.

   To ensure the multi-dimensional aspects of chronic pain experienced by individuals are measured adequately, pain assessment tools have been selected that will address different aspects of each participant's' chronic pain and functional capacity. To measure the impact of VR on each participant's pain intensity, the Visual Analog Scale will be used during the VR and control experiences, pre and post exposure and at 10 minute intervals. In order to measure the change in pain during the therapy experience, and overall sleep quality, at the end of each week, participants will also be asked to complete post-intervention questionnaires: Health Survey (Short-Form 12), McGill Pain Questionnaire, the Pittsburgh Sleep Quality Index, and also a brief Virtual Reality Immersion Tool (to assess how immersive they found the experience that week).
2. Interpretive Description Study (Qualitative):

A Qualitative Interpretative-Descriptive exploration will be undertaken alongside the trial to allow for a more open exploration of participants experiences and to further understanding of the perceptions associated with the use of immersive multimedia and any impact upon their chronic pain. An interpretative description (ID) approach will be used for this aspect of the study. This methodology allows for an inductive descriptive analysis of the phenomena, and was chosen as it is ideal for small scale studies, allowing for generation of themes, patterns and theory associated with the patient's experience.

Following the completion of the clinical trial all participants will be sent an exploratory questionnaire to discover their perceptions of immersive multimedia and its value (if any) in the control of their chronic pain. In this questionnaire they will also be invited to participate in one of two focus group interviews. Data from this will be analyzed and used to support purposeful sampling of individuals to take part in the following focus-group interviews, to include those subjects with a range of diverse opinions and ideas. As themes and categories emerge from the data the researchers will seek to adapt the focus-group interview sample with the purpose of strengthening the emerging theory and patterns by including individuals who will help further define the characteristics of these themes and categories.

Data Analysis

Quantitative Data: Descriptive and inferential statistical analysis will be performed on the pain scores. For face-value quantitative indicators of potential effects univariate descriptive statistics will be employed. Data will be analyzed for central tendency, dispersion (standard deviation, interquartile range), skewness and kurtosis using SPSS statistical analysis software to establish distribution and variance. Likewise, quantitative data from the questionnaires will be analysed in this fashion. Data will be explored for differences in the pain scales for the VR group and the control group at each time point to analyze for any indications of changes immediately following the experience using Linear Mixed Effects Modelling using SPSS software.

Qualitative Data: The focus-group interviews will be audiotaped. The questionnaire open text results and transcriptions of focus groups will be recorded into NVivo 11.0 qualitative data analysis software and read, re-read and coded for thematic elements by the PIs.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or older
* Previous or current medical diagnosis of cancer
* Previous or current treatment by chemotherapy, radiotherapy, hormonal
* Currently an outpatient (not hospitalized)
* Chronic pain sufferer (suffering ongoing daily pain for 3 months or more with a Neuropathic Rating Pain Scale score of 4 or more)
* Able to understand the English language, and read and write English
* Have normal stereoscopic (binocular) vision
* Able to easily move your head up, down, left and right and wear a headset
* Have fine motor control in one hand sufficient to operate a joystick/control
* Have space at home for a computer and monitor equipment

Exclusion Criteria:

* Cognitive impairment/inability to control a basic computer VR interface, or complete questionnaires
* Receiving regular non-pharmacological pain relieving adjunct therapies for the management of chronic pain
* Susceptibility to motion sickness/cyber-sickness
* Susceptibility to claustrophobia (fear of confined places)
* History of susceptibility to seizures

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard M Garrett, Ph.D., Principal Investigator — University of British Columbia - School of Nursing
Locations (3):
- Canada (3):
  - Simon Fraser University - School of Interactive Arts and Technology, Surrey, British Columbia
  - University of British Columbia - School of Nursing, Vancouver, British Columbia
  - BC Cancer, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
We can share the study protocol, statistical analysis plan, informed consent form as well as the analytic code used.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Please reach out to us. Data will be available for a year after the study concludes.
Access Criteria: Connect with researcher.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a parallel two-arm (VR vs non-VR control) participant blinded prospective RCT with 1:1 allocation. It was primarily conducted with rolling recruitment in British Columbia as well as Alberta, Ontario and Quebec between August 2017 and December 2022. Participants were given either all the equipment necessary to complete the study in their homes.
Pre-assignment Details: Interested participants were screened for eligibility and assigned a participant ID by the research coordinator. The research assistant responsible for equipment setup would then determine the participant's group from the assignment sheet. Participants were randomly assigned to either the VR or control group in blocks of 12 using a Latin Square design assignment sheet prepared by a professional statistician.
Groups:
- VR Group (Intervention Group): Participants were randomly assigned to the intervention group. The VR interventions are identical for each participant and consist of a PC running the immersive virtual reality application with a Virtual Reality headset that allows for 110 degrees field of view. The interventions are one month in length to enable customization to the therapy and record data over a long enough period of time to account for individual short-term changes in pain experience. Participants used the VR interventions every day with a time exposure of 30 minutes for four consecutive weeks. There was one rest day a week (normally a Sunday) where no therapy is given.
  The following VR experiences were used in the VR group:
  Virtual Meditative Walk: http://painstudieslab.com/projects/virtual-meditative-walk/ Wildflowers: https://appadvice.com/app/wildflowers-mindfulness/988835763 Obduction: http://obduction.com/ Carpe Lucem: http://store.steampowered.com/app/433700/Carpe_Lucem__Seize_The_Light_VR/
- 2D Computer Group (Control Group): Participants were randomly assigned to the control group. The control group applications were identical for each participant. The control group was exposed to 2D PC equivalent versions of the same multimedia experiences but on their PC screen (without the Virtual Reality headset use). These are functionally similar to the VR experiences. Participants used the applications every day with a time exposure of 30 minutes for four consecutive weeks. There was one rest day a week (normally a Sunday) where no application is given.
  The following PC applications were used in the control group:
  Virtual Meditative Walk: http://painstudieslab.com/projects/virtual-meditative-walk/ Wildflowers: https://appadvice.com/app/wildflowers-mindfulness/988835763 Obduction: http://obduction.com/ The Witness: http://store.steampowered.com/app/210970/
Period: Overall Study
Arm/Group | VR Group (Intervention Group) | 2D Computer Group (Control Group)
Started | 57 | 53
Completed | 50 | 50
Not Completed | 7 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 6 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is not different from the assignment population.
Groups:
- Intervention Group: Participants were randomly assigned to the intervention group. The VR applications are identical for each participant and consist of a PC running the immersive virtual reality application with a Virtual Reality headset that allows for 110 degrees field of view. The applications are one month in length to enable customization to the therapy and record data over a long enough period of time to account for individual short-term changes in pain experience. Participants used the VR applications every day with a time exposure of 30 minutes for four consecutive weeks. There was one rest day a week (normally a Sunday) where no applications is used.
  The following VR applications were used in the VR group:
  Virtual Meditative Walk: http://painstudieslab.com/projects/virtual-meditative-walk/ Wildflowers: https://appadvice.com/app/wildflowers-mindfulness/988835763 Obduction: http://obduction.com/ Carpe Lucem: http://store.steampowered.com/app/433700/Carpe_Lucem__Seize_The_Light_VR/
- Control Group: Participants were randomly assigned to the control group. The control group applications were identical for each participant. The control group was exposed to 2D PC equivalent versions of the same multimedia experiences but on their PC screen (without the Virtual Reality headset use). These are functionally similar to the VR experiences. Participants used the applications every day with a time exposure of 30 minutes for four consecutive weeks. There was one rest day a week (normally a Sunday) where no application is given.
  The following PC applications were used in the control group:
  Virtual Meditative Walk: http://painstudieslab.com/projects/virtual-meditative-walk/ Wildflowers: https://appadvice.com/app/wildflowers-mindfulness/988835763 Obduction: http://obduction.com/ The Witness: http://store.steampowered.com/app/210970/
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (13.5) | 58.3 (10.2) | 56.9 (12.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 16 | 14 | 30
  Not Disclosed | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 50 | 50 | 100
Visual Analog Pain Scale (VAS) [Mean (Full Range); unit: units on a scale] — The Visual Analog Scale (VAS) is a psychometric tool used to measure the subjective characteristics of perceived pain are difficult to measure directly.
  Collected as a baseline measure and weekly thereafter for 4 weeks.
  units on a scale | 5.0 [0 to 10] | 4.4 [0 to 10] | 4.7 [0 to 10]
Short Form McGill Pain Questionnaire (SF-MPQ) [Mean (Full Range); unit: units on a scale] — The short-form McGill Pain Questionnaire is a standardized qualitative pain assessment tool that was created to assess both the intensity and quality of pain.
  Collected as a baseline measure and weekly thereafter for 4 weeks.
  units on a scale | 22 [0 to 78] | 24 [0 to 78] | 23 [0 to 78]

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS)
Description: Daily pain was assessed using the Visual Analogue Scale (VAS). The VAS is a single item linear self-reported pain scale from no pain (0mm) to worst pain imaginable (100mm). The clinically meaningful change for the VAS has been shown to be between 9mm and 12mm; for this study adopted the convention of 10mm as the minimum clinically important difference (MCID).
Time Frame: Right before intervention (Pre), during intervention (During) and right after intervention (Post)
Population: Participants with pain scores before, during and after each immersion session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | VR Group (Intervention Group) | 2D Computer Group (Control Group)
Number analyzed (Participants) | 49 | 48
units on a scale
  Pre to During | -9.64 (0.63) | -7.56 (0.63)
  Pre to Post | -7.91 (0.63) | -8.43 (0.63)
Statistical Analysis 1: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Null hypothesis: There is no difference between the reported daily pain experiences of participants during, or after exposure to VR immersive environments, overall and within four different VR immersive environments, compared to the equivalent applications experienced on a 2D computer screen; Test type: Equivalence — As reliable estimates of expected effect size were unknown, the study was powered to detect a medium effect (0.5 SD change), considered a reasonable clinically meaningful impact to obtain 80% power based on a repeated measures analysis of variance (RM ANOVA) with 2-tailed alpha of .05 model; Mean Difference (Net) = -2.08, 95% CI 2-sided [-3.86 to -0.30] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 2: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.53, 95% CI 2-sided [-1.24 to 2.37] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method

2. Secondary Outcome: McGill Pain Questionnaire
Description: The McGill Pain Questionnaire (MPQ) is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is a dimensional tool for pain assessment and it has three components, which are the sensory intensity, the cognitive evaluation of pain and the emotional impact of pain. The MPQ is composed of 78 words, of which respondents choose those that best describe their experience of pain. Seven words are selected from the following categories: dimension 1 to 10 (pain descriptors), three words; dimensions 11 to 15 (affective components of pain), dimension 16 (evaluation of pain) one word, and dimension 17 to 20 (miscellaneous) one word. Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain). Qualitative differences in pain may be reflected in respondent's word choice.
Time Frame: Before the start of the weekly VR session and after the weekly VR session for a period of 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | VR Group (Intervention Group) | 2D Computer Group (Control Group)
Number analyzed (Participants) | 50 | 50
units on a scale
  Change in score at week 1 from baseline | -0.90 (1.04) | -1.98 (1.03)
  Change in score at week 2 from baseline | -2.02 (1.04) | -4.48 (1.03)
  Change in score at week 3 from baseline | -3.36 (1.05) | -3.75 (1.04)
  Change in score at week 4 from baseline | 2.88 (1.05) | -5.44 (1.03)
Statistical Analysis 1: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See section for primary outcome; Mean Difference (Net) = 1.08, 95% CI 2-sided [-1.59 to 3.95] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 2: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See section on primary outcome; Mean Difference (Net) = 2.16, 95% CI 2-sided [-0.55 to 5.08] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 3: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See section on primary outcome; Mean Difference (Net) = 0.39, 95% CI 2-sided [-2.64 to 3.42] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 4: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See section on primary outcome; Mean Difference (Net) = 2.56, 95% CI 2-sided [-0.08 to 5.48] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method

3. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: the Pittsburgh Sleep Quality Index (PSQI) was used as a self-reported outcome measure assessing sleep quality at the end of each week. The measure includes 19 items asking about sleep schedule, duration, disruption frequency (4-point Likert scale), and quality (4-point Likert scale) using worse 0 to best 3. Scores are summed and range from 0-21, with higher scores indicating worse sleep quality.
Time Frame: Before the start of the weekly VR session and after the weekly VR session for a period of 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Intervention Group: Participants will be randomly assigned to the intervention group (50 in total).The VR intervention will be identical for each participant and consist of a PC running the immersive virtual reality application with a Virtual Reality headset 110 degrees field of view head mounted display. The VR will be a set of commercial exploratory virtual environment games designed for the HTC Vive headset. The intervention will be used for one month to enable customization to the therapy and record data over a long enough period of time to account for individual short- term changes in pain experience. Participants will be asked to use the VR therapy every day with a time exposure of 30 minutes for four consecutive weeks. There will be one rest day a week (normally a Sunday) where no therapy is given.
  Virtual Reality Headset: The following VR experiences will be used:
  Virtual Meditative Walk: http://painstudieslab.com/projects/virtual-meditative-walk/ Wildflowers: https://appadvice.com/app/wildflowers-mindfulness/988835763 Obduction: http://obduction.com/ Carpe Lucem: http://store.steampowered.com/app/433700/Carpe_Lucem__Seize_The_Light_VR/
- Control Group: The control group will be exposed to 2D PC equivalent versions of the same multimedia experiences but on their PC screen (without the Virtual Reality headset use). These will be functionally similar to the VR experiences.
  2D PC: The control group will be exposed to 2D equivalent versions of the same multimedia experiences but on their PC screen (without the VR headset use). These will be functionally similar to the VR experiences. These will include:
  Virtual Meditative Walk: http://painstudieslab.com/projects/virtual-meditative-walk/ Wildflowers: https://appadvice.com/app/wildflowers-mindfulness/988835763 Obduction: http://obduction.com/ The Witness: http://store.steampowered.com/app/210970/
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 50 | 50
units on a scale
  Change at week one from baseline | -0.13 (0.41) | 0.50 (0.41)
  Change at week two from baseline | -0.24 (0.42) | -0.86 (0.42)
  Change at week three from baseline | -0.84 (0.41) | -0.71 (0.42)
  Change at week four from baseline | -0.94 (0.42) | -1.26 (0.41)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = 0.37, 95% CI 2-sided [-0.71 to 1.5] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = 0.62, 95% CI 2-sided [-0.49 to 1.89] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Test type: Equivalence — See comments in primary outcome; Mean Difference (Net) = -0.13, 95% CI 2-sided [-1.19 to 1.09] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 4: Comparison: Intervention Group vs Control Group; Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = 0.33, 95% CI 2-sided [-0.88 to 1.57] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method

4. Secondary Outcome: 12 Item Short Form Health Survey (SF-12) Physical Health Component Score
Description: The SF-12 is used to assess the impact of health on an individual's everyday life over the 4 weeks interval. It includes 12 items with binary response items (yes/no) and 3-6-point Likert items (worse to best). The SF-12 is scored using proprietary software to generate a physical composite (PCS) and mental composite (MCS) health scores ranged 0-100, with scores above or below 50 indicating greater or poorer health than the normative mean, respectively.
Time Frame: Before the start of the weekly VR session and after the weekly VR session for a period of 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | VR Group (Intervention Group) | 2D Computer Group (Control Group)
Number analyzed (Participants) | 50 | 50
units on a scale
  Change in score at week one from baseline | 2.03 (0.92) | -0.45 (0.93)
  Change in score at week two from baseline | 1.38 (0.92) | -0.66 (0.93)
  Change in score at week three from baseline | 3.40 (0.92) | -0.39 (0.94)
  Change in score at week four from baseline | 2.80 (0.92) | -0.38 (0.92)
Statistical Analysis 1: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = 2.48, 95% CI 2-sided [0.02 to 4.70] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 2: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = 2.04, 95% CI 2-sided [-0.42 to 4.39] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 3: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = 3.79, 95% CI 2-sided [1.02 to 6.08] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 4: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = 3.18, 95% CI 2-sided [0.68 to 5.69] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method

5. Secondary Outcome: 12 Item Short Form Health Survey (SF-12) Mental Health Component Score
Description: The SF-12 is used to assess the impact of health on an individual's everyday life over the 4 weeks interval. It includes 12 items with binary response items (yes/no) and 3-6-point Likert items. The SF-12 is scored using proprietary software to generate a physical composite (PCS) and mental composite (MCS) health scores ranged 0-100, with scores above or below 50 indicating greater or poorer health than the normative mean, respectively.
Time Frame: Before the start of the weekly VR session and after the weekly VR session for a period of 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | VR Group (Intervention Group) | 2D Computer Group (Control Group)
Number analyzed (Participants) | 50 | 50
units on a scale
  Change in score at week one from baseline | 0.68 (1.19) | 2.99 (1.20)
  Change in score at week two from baseline | 0.37 (1.19) | 4.27 (1.20)
  Change in score at week three from baseline | 1.51 (1.19) | 2.38 (1.21)
  Change in score at week four from baseline | 2.27 (1.19) | 5.22 (1.20)
Statistical Analysis 1: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = -2.31, 95% CI 2-sided [-5.63 to 0.98] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 2: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = -3.90, 95% CI 2-sided [-7.35 to -0.48] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 3: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See comment in primary outcome; Mean Difference (Net) = -0.87, 95% CI 2-sided [-4.11 to 2.62] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method
Statistical Analysis 4: Comparison: VR Group (Intervention Group) vs 2D Computer Group (Control Group); Test type: Equivalence — See comments in primary outcome; Median Difference (Net) = -2.95, 95% CI 2-sided [-6.10 to 0.41] — Treatment effect = VR group - Control group; 95% confidence intervals estimated using the bootstrapping method

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the entirety of the trial participation (up to 4 weeks) from the initial baseline recording of data to the end of the participants use of the multimedia/VR equipment. They were not recorded after participants ceased use of the equipment. Cybersickness self-reporting was undertaken every week during use of the equipment on a weekly basis. Participants were asked to report any events of sickness during the preceding week on a Friday.
Description: The use of VR and 2D laptop computers have been established as clinically safe and are commonly used recreationally. VR users were screened for risk of epilepsy, seizures and motion sickness during recruitment as exclusion criteria to prevent participation of those at increased risk of those adverse events.
Arm/Group | VR Group (Intervention Group) | 2D Computer Group (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 35/50 | 8/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VR Group (Intervention Group) (N=50) | 2D Computer Group (Control Group) (N=50)
Cybersickness (General disorders) | 35 (61) | 8 (16) — Cybersickness is a form of motion sickness that occurs as a result of exposure to immersive environments, such as virtual reality (VR) and augmented reality (AR) applications.

LIMITATIONS AND CAVEATS:
There were several imitations in this study. First, the external validity may be limited as the types of cancer patients participating and pain types were heterogenous, and participant self-selection may mean they were not representative of the larger cancer chronic pain population. Secondly, the study may have been statistically underpowered due to the effect size selected, intervention exposure time, and multiple VR applications used as dependent variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT02995434/Prot_SAP_000.pdf